CLINICAL TRIAL: NCT06064058
Title: Assessing the Effects of HbA1c Reduction on Alleviating Nonspecific Back Pain in Prediabetic Non-obese Patients: A Randomized Controlled Trial
Brief Title: Assessing the Effects of HbA1c Reduction on Alleviating Nonspecific Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Doctor (MBChB), University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2023-09-24; First posted 2023-10-03 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Back Pain Lower Back Chronic; Back Pain; Pre Diabetes; Diabetes; Back Pain, Low
Keywords: Back Pain; HBA1C
MeSH Terms: conditions — Back Pain; Glucose Intolerance; Diabetes Mellitus; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Three Groups:
  * Case
  * Palcebo
  * No placebo, no intervention group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interventional group (Experimental): This group were assigned to 6-month lifestyle modification program, focusing on diet, sleep, exercise, and vitamin D and magnesium correction.
  Interventions: Dietary Supplement: Ghazwan program
- Control group (Placebo Comparator): Ordinary painkillers given
  Interventions: Drug: Standard management
- No Placebo, no intervention group (No Intervention): Nothing was given to them neither 6-month lifestyle modification program, focusing on diet, sleep, exercise, and vitamin D and magnesium correction nor painkillers.

INTERVENTIONS:
Dietary Supplement: Ghazwan program — 6-month lifestyle modification program, focusing on diet, sleep, exercise, and vitamin D and magnesium correction.
  Arms: Interventional group
Drug: Standard management — Standard care with NSAIDs and acetaminophen for pain management
  Arms: Control group

SUMMARY:
Prediabetes, characterized by elevated HbA1c levels, is a common precursor to type 2 diabetes mellitus. Recent studies have suggested a potential link between prediabetes and nonspecific back pain. This randomized controlled trial aimed to assess whether reducing HbA1c levels through lifestyle interventions and, along with the correction of vitamin D and magnesium, can alleviate nonspecific back pain in prediabetic patients.

DETAILED DESCRIPTION:
The study included 40 patients from an outpatient clinic in Baghdad, evenly divided into intervention and control groups. The intervention group underwent a 6-month lifestyle modification program, focusing on diet, sleep, exercise, and vitamin D and magnesium correction. HbA1c levels were measured, and back pain severity was assessed (through what assessment method ?). The control group received standard care with NSAIDs and acetaminophen for pain management. Assessments were conducted at baseline and at various intervals over a total period of 6 months to evaluate changes in HbA1c levels and back pain intensity.

This randomized controlled trial provides evidence that reducing HbA1c levels through lifestyle modifications, along with the correction of vitamin D and magnesium, can lead to a reduction in nonspecific back pain intensity and improved functional outcomes in prediabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Poor sleep (less than 6 hours per day)
* chronic back pain
* Multiple joint pain
* non-specific back pain
* HBA1C more than 5.7
* ability to record the data

Exclusion Criteria:

* Not able to record data
* previous spine surgeries
* severe OA in knee
* Spinal stenosis
* Peripheral vascular diseases
* Rheumatological diseases
* Lumbar disc prolapse
* uncooperative patient

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
HBA1C | 6 months
  Diabetes index

CONTACTS AND LOCATIONS:
Overall Officials: Hashim T Hashim, MBChB, Study Director — University of Warith Al-Anbiyaa, College of Medicine
Locations (1):
- Dr. Ghazwan A. Hasan Clinic, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No